CLINICAL TRIAL: NCT01066156
Title: Functional Reciprocity Between Heightened Stress Reactivity and Emotional Numbing in PTSD: Novel Predictors of Pharmacotherapeutic Outcomes
Brief Title: Post-Traumatic Stress Disorder (PTSD) and Seroquel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge Health Alliance (Other)
Responsible Party: Principal Investigator, Igor Elman, MD, Cambridge Health Alliance
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-P-001664
Record Dates: First submitted 2010-02-08; First posted 2010-02-10 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2015-06

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: Post-traumatic Stress Disorder; PTSD; Seroquel; fMRI
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Seroquel (Experimental): This study will investigate therapeutic responses to Seroquel pharmacotherapy in PTSD
  Interventions: Drug: Seroquel

INTERVENTIONS:
Drug: Seroquel — This study will investigate therapeutic responses to Seroquel pharmacotherapy in PTSD
  Other Names: quetiapine

SUMMARY:
This 8 weeks study will investigate therapeutic responses to Seroquel pharmacotherapy in PTSD.

DETAILED DESCRIPTION:
An initial telephone interview will be conducted to determine if potential subjects meet the basic study requirements. If no obvious counterindications are present, subjects will be scheduled for a screening visit. After briefing the subjects on the reasons for the research, they will be given an opportunity to read the Informed Consent Form, approved by the Cambridge Health Alliance Institutional ReviewBoard, and to ask questions prior to signing it. Subjects will be given a copy of the signed Consent Form. Each subject will complete a standardized interview schedule designed to obtain personal and background data along with psychodiagnostic and psychometric evaluations. An open-label treatment will be utilized for all patients. Seroquel tablets will be flexibly dosed and begun at a target dose of 25 mg per day and taken over an 8 week period.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Fluency in English
* A diagnosis of PTSD
* No pregnancy
* Right-handedness

Exclusion Criteria:

* Pregnancy or lactation
* Any cognitive impairment that precludes informed consent
* Known intolerance or lack of response to Seroquel
* Previous enrollment or randomization of treatment in the present study
* Participation in another drug trial within 4 weeks prior enrollment into this study
* Patients with Diabetes Mellitus
* History of allergic reaction or hypersensitivity to Seroquel
* Contraindications to magnetic resonance imaging
* Treatment with an effective medication for PTSD

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Igor Elman, MD, Principal Investigator — CHA
Locations (1):
- Central Street Health Center, Somerville, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Seroquel
Started | 34
Completed | 24
Not Completed | 10
Not completed — ineligible | 2
Not completed — Lost to Follow-up | 7
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Seroquel
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 34
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 18
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in PTSD Symptomatology at the Week 8 Timepoint.
Description: We will compare patients' symptomatology at baseline vs. at 8 week timepoint
  Specify Full Scale Name and Construct (i.e., indicate what the scale measures if not clear from name): Clinician-Administered PTSD Scale (CAPS)
  Include all scale ranges (i.e., minimum and maximum scores) required to interpret any values in the data table: 0-136
  For each scale range provided, specify which values are considered to be a better or worse outcome: 0-best, 136 worst
  If subscales are combined to compute a total score, consider indicating how subscales are combined (summed, averaged, etc.): summed
Time Frame: 8 weeks
Population: It was predicted that patients will show a change in PTSD symptoms as measured by the Clinician Administered PTSD Scale (CAPS).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Seroquel
Number analyzed (Participants) | 24
units on a scale | 7.3 (18.5)

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Seroquel
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes